CLINICAL TRIAL: NCT00005712
Title: Self Management Education Asthma
Status: Terminated | Type: Observational
Why Stopped: Not a clinical trial and was inadvertently entered in the system.
Sponsor: University of New Mexico (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4921; R01HL045279 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To evaluate the effects of a new statewide program to enhance identification, referral and provision of care to rural families of Hispanic children with moderately severe to severe asthma. Specifically, to determine if comprehensive medical care (CMC) plus an educational self-management program for rural Hispanic children and their families had an impact on asthma morbidity, as well as on cost and family adaptation.

DETAILED DESCRIPTION:
BACKGROUND:

Because of New Mexico's large rural and heavily Hispanic population, it was an ideal setting to determine effective methods for case management, self-management educational programs and effective tertiary to primary care delivery collaboration.

The study was part of a demonstration and education initiative "Interventions for Control of Asthma Among Black and Hispanic Children" which was released by the NHLBI in June 1989.

DESIGN NARRATIVE:

A randomized block design was used with random assignment of subjects by county to treatment groups of 1. comprehensive medical care or standard tertiary care and education, or 2. CMC-Plus adding a structured self-management program--Open Airways/Respiro Abierto (developed and tested with support of NHLBI). CMC-Plus also received in home education and intervention from community based Hispanic family educators trained in an empowerment model of family intervention, in-home support, and education. Case management was provided by CMS; CMC and CMC-Plus were provided at the UNM-PPP in close collaboration with and transfer of care to the primary physician. Additional educational contact with primary care providers and emergency rooms were provided through the UNM Department of Family, Community & Emergency Medicine which utilized the National Institutes of Health National Asthma Education Program's Guidelines for Step-Wise Care of Asthma. Asthma morbidity, cost of care, family adaptation and family satisfaction were evaluated using standardized instruments.

ELIGIBILITY:
No eligibility criteria

Ages: 0 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-08; Study Completion 1996-07

REFERENCES:
- [Background] Clark D, Gollub R, Green WF, Harvey N, Murphy SJ, Samet JM. Asthma in Jemez Pueblo schoolchildren. Am J Respir Crit Care Med. 1995 May;151(5):1625-7. doi: 10.1164/ajrccm.151.5.7735623.